CLINICAL TRIAL: NCT03067051
Title: Open-label Clinical Study to Assess the Safety and Efficacy of the SpectraCure P18 System (Interstitial Multiple Diode Lasers and IDOSE® Software) and Verteporfin for Injection (VFI) for the Treatment of Recurrent Prostate Cancer
Brief Title: Clinical Study to Assess the Safety and Efficacy of the SpectraCure P18 System
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SpectraCure AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPC11-01-110
Record Dates: First submitted 2017-02-13; First posted 2017-03-01 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Verteporfin

STUDY DESIGN:
Intervention Model Description: As result of the accelerated titration design with light dose and verteporfin for injection (VFI), the final number of subjects depends on the outcome of the titration. If all dose levels enroll and complete at the minimum number of subjects, the number of subjects is 12 (1 each at dose levels 1-3, 3 each at dose levels 4-6). If all dose levels enroll and complete at the maximum number of subjects, the number of subjects is 36 (6 subjects at each dose level 1-6). The range is thus 12-36 subjects for the dose-escalation phase.
  25-30 subjects will be treated in an expanded cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- PDT and verteporfin dose finding (Experimental): Verteporfin and Interstitial Photodynamic Therapy are the interventions in this dose titration study.
  The interventions will be light dose (as laser) using the SpectraCure P18 System and drug intervention with verteporfin as a photosensitizer.
  The study will be conducted as a dose titration study to determine the light and drug threshold dose using the SpectraCure P18 System (Interstitial multiple diode lasers and IDOSE® Software) and verteporfin for injection (VFI).
  The light is delivered to the tumor via optical fibers and each dose arm will receive Interventional Photodynamic Therapy of Prostate Cancer combined with the drug verteporfin as a photosensitizer .
  Interventions: Drug: Verteporfin; Device: SpectraCure P18 System

INTERVENTIONS:
Drug: Verteporfin — In the last decade a clinical interest of developing new methods for minimally invasive treatments of organ-confined prostatic malignancies has been pursued. In this study the drug verteporfin for injection (VFI) is to be used with the SpectraCure P18 System (Interstitial multiple diode lasers and IDOSE® Software).
  Other Names: Visudyne
Device: SpectraCure P18 System — Interstitial Photodynamic therapy is provided with the the SpectraCure P18 system

SUMMARY:
The rationale for the study is to obtain safety and efficacy data as well as to establish dose parameters for the SpectraCure P18 System with IDOSE®, with verteporfin for injection (VFI) as photosensitizer for the treatment of recurrent prostate cancer.

DETAILED DESCRIPTION:
In 2011, more than 200,000 men in North America alone were diagnosed with cancer of the prostate, which makes it one of the most common cancer types. It affects the lives of the subjects in many ways.

After treatment the subjects PSA levels are being closely monitored to detect potential recurrence. A high number of subjects will get recurrent prostate cancer. The treatment options for recurrent cancer are more limited than for primary tumors as secondary treatment partly depends on which treatment the subject has previously undergone.

Treatment of recurrent prostate cancer may, depending on the standard treatment of the primary disease, include the following:

* Radiation therapy.
* Prostatectomy for subjects initially treated with radiation therapy.
* Hormone therapy.
* Pain medication, external radiation therapy, internal radiation therapy with radioisotopes such as strontium-89, or other treatments as palliative therapy to lessen bone pain.

The objectives of this study is to demonstrate that the use of the SpectraCure P18 System (Interstitial multiple diode lasers and IDOSE® Software) and verteporfin for injection (VFI) is a safe treatment for recurrent prostate cancer.

ELIGIBILITY:
Phase 1 Inclusion Criteria:

1. Males > 18 years who have gone through external or internal, high dose rate (brachy) radiation therapy for localized prostate cancer with histopathologically verified local recurrence.
2. Prostate volume less than 50 cm3 defined by transrectal ultrasound
3. Subject not eligible for surgery or curative radiotherapy
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Expected survival ≥ 8 months
6. Sufficient bone marrow reserve as indicated by; granulocyte count ≥ 1500/mm3, platelet count ≥ 100,000/mm3
7. Adequate renal function as defined by creatinine ≤ 1.5 mg /dl
8. Adequate hepatic function, based on a total bilirubin ≤ 1.5 mg/dl, serum glutamate-oxaloacetate transaminase (SGOT) ≤ 3 times the upper limit of normal, and alanine transaminase (ALT) ≤ 3 times the upper limit of normal
9. Signed Informed Consent

Phase 1 Exclusion Criteria:

1. Patients with locally advanced (AJCC 7th edition T3/T4) or metastatic disease
2. Patients who have been treated with seed implantation brachytherapy
3. Gleason score ≥ 8 at initial diagnosis
4. Less than 1 week since surgery (excluding minimal procedures, e.g. vascular access device insertion)
5. Concomitant infection
6. Subjects with other severe concurrent disease that in the judgement of the investigator would make the subject inappropriate for entry into this study
7. Mental incapacity or psychiatric illness that would interfere with the subject's ability to understand and give informed consent or to complete follow-up visits according to the judgement of the investigator
8. Contraindication for photosensitizer
9. Porphyria or other diseases exacerbated by light
10. Known hypersensitivity to verteporfin for injection (VFI) or to any of the excipients
11. Known allergies to porphyrins
12. Tumours known to be eroding into a major blood vessel in or adjacent to the illumination site
13. On-going therapy with a photosensitizing agent
14. Enrolment in another therapeutic clinical study within 3 months prior to randomization and throughout the study.
15. Subjects with a history of CTCAE v4 grade 3 or greater or persistent (>1 separate episode or symptoms lasting more than 3 months after initiation of medical intervention) grade 2 proctitis attributed to radiation.

Phase 2 Inclusion Criteria:

1. Subjects > 18 years who have gone through external or internal, high dose-rate (brachy) radiation therapy for localized prostate cancer with histopathologically verified local recurrence.
2. Treatment target volume less than 50 cm3.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Expected survival ≥ 12 months.
5. Sufficient bone marrow reserve as indicated by; granulocyte count ≥ 1500/mm3, platelet count ≥ 100,000/mm3.
6. Adequate renal function as defined by creatinine ≤ 1.5 mg /dl.
7. Adequate hepatic function, based on a total bilirubin ≤ 1.5 mg/dl, serum glutamate- oxaloacetate transaminase (SGOT) ≤ 3 times the upper limit of normal, and alanine transaminase (ALT) ≤ 3 times the upper limit of normal.
8. Signed Informed Consent.

Phase 2 Exclusion Criteria:

1. Subjects with locally advanced (AJCC 7th edition T3/T4), regional pelvic lymph node metastasis, or metastatic disease defined by PSMA PET.
2. Subjects who have been treated with seed implantation brachytherapy.
3. Less than 1 week since surgery (excluding minimal procedures, e.g. vascular access device insertion).
4. Concomitant infection.
5. Subjects with other severe concurrent disease that in the judgement of the investigator would make the subject inappropriate for entry into this study.
6. Mental incapacity or psychiatric illness that would interfere with the subject's ability to understand and give informed consent or to complete follow-up visits according to the judgement of the investigator.
7. Contraindication for photosensitizer.
8. Porphyria or other diseases exacerbated by light.
9. Known hypersensitivity to verteporfin for injection (VFI) or to any of the excipients.
10. Known allergies to porphyrins.
11. Tumours known to be eroding into a major blood vessel in or adjacent to the illumination site.
12. On-going therapy with a photosensitizing agent.
13. Enrolment in another therapeutic clinical study within 3 months prior to randomization and throughout the study.
14. Subjects with a history of CTCAE v4 grade 3 or greater or persistent (>1 separate episode or symptoms lasting more than 3 months after initiation of medical intervention) grade 2 proctitis attributed to radiation.
15. Contraindication for MRI/Gadolinium contrast such as: implants, severe renal impairment (glomerular filtration rate [GFR] <30 mL/min/1.73m2, or previous contrast reactions.
16. On-going or planned hormone therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with recurrent prostate cancer
Enrollment: 66 (Estimated)
Dates: Start 2017-03-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assesses by CTCAE v4.0 related to protocol therapy. | Within 4 weeks of treatment in each cohort.
  Dose limiting toxicities are defined as grade 3 non-hematologic or grade 4 hematologic toxicities that are possibly, probably or definitely related to PDT.
Percentage of subjects with negative biopsies. | 6 months following PDT.
  Histopathologically tumor-free.

SECONDARY OUTCOMES:
Damage to the periprostatic tissues including the rectal wall mediated by PDT | 5-9 days following PDT
  Potential damage to the periprostatic tissue will be evaluated by contrast-enhanced and not-contrast enhanced MRI.
Performance of SpectraCure P18 system | Dose-volume histograms will be evaluated at month 12
  Performance of the SpectraCure P18 system will be evaluated by light dose-volume histograms for the light dose coverage
Adequacy of effectiveness | Within 1 week of treatment
  Effectivity will be evaluated by MRI to determine the extent of necrosis in the prostate
Percentage of subjects with remaining localized tumour. | 12 months following PDT.
  Evaluated by MRI.
Percentage of subjects with biochemical failure. | 12 months following PDT.
  Failure defined as a rise in PSA level of 2.0 ng/mL or more, over and above the nadir.
Percentage of subjects with extra prostatic or distant disease. | 12 months following PDT.
  Evaluated by PSMA PET.

CONTACTS AND LOCATIONS:
Locations (4):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Skåne University Hospital, Malmo, Skåne County, Sweden
- Reader in Urology, University College London & Honorary Consultant Urological Surgeon, University College London Hospitals Trust, London, United Kingdom